CLINICAL TRIAL: NCT06643650
Title: PHASE IV Observational Study to Document the Phenomenon of Vitamin D Deficiency and Its Added Value in Patients with Low-energy Osteoporotic Hip Fracture, in Daily Practice in Greece.
Brief Title: Study to Document the Phenomenon of Vitamin D Deficiency and Its Added Value in Patients with Low-energy Osteoporotic Hip Fracture, in Daily Practice in Greece.
Status: Recruiting | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, EFSTATHIOS CHRONOPOULOS, Professor of Orthopaedic Surgery, National and Kapodistrian University of Athens
Other Study IDs: 945/11-03-2022
Record Dates: First submitted 2024-02-07; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-02

CONDITIONS: Vitamin D Deficiency; Osteoporosis; Bone Loss, Age-Related; Fracture of Hip
MeSH Terms: conditions — Vitamin D Deficiency; Osteoporosis; Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 1st group: 3 months intake of cholecalciferol supplementation (therapeutic dose)
  Interventions: Dietary Supplement: CHOLECALCIFEROL ORAL.SOL 25000 IU/2,5ML
- 2nd group: 3 months therapeutic and 3 months prophylactic dose intake of cholecalciferol
  Interventions: Dietary Supplement: CHOLECALCIFEROL ORAL.SOL 25000 IU/2,5ML

INTERVENTIONS:
Dietary Supplement: CHOLECALCIFEROL ORAL.SOL 25000 IU/2,5ML — Cholecalciferol 25000IU/week for 3 months in both groups. 2nd group continues with 25000IU/month for following 3 months.
  Other Names: DELTIUS ORAL.SOL 25000 IU/2,5ML

SUMMARY:
Vitamin D, through its action on calcium metabolism, is essential for bone physiology. Vitamin D deficiency can affect muscle function and increase the risk of falls in the elderly, while severe deficiency is common in patients with fragility fractures. Vitamin D and calcium supplementation, in addition to anti-osteoporosis treatment after surgery or conservative treatment, can ensure optimal recovery and survival, especially in patients with a hip fracture.

The goal of vitamin D supplementation is to bring the serum 25-(OH)-D concentration above 30 ng/ml.

Clinical pathways have been developed to support orthopedic surgeons in improving the medical management of patients after orthopedic/surgical fracture management. Pathways include advising primary care physicians and orthopedic surgeons on diagnostic and therapeutic approaches, promoting their appropriate use without compromising quality of care, and educating patients on non-pharmacological management of their disease (physical therapy, lifestyle habits life and nutrition).

This is an observational cohort study that will record data on the use of vitamin D in daily practice in patients with low-energy fractures.

The aim of this study is to measure vitamin D levels in the patient and provide these patients according to daily practice with appropriate supplementation for a period of one year, observing if there is a good functional outcome and a reduction in the risks of new fractures.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old
* Patients with a low energy fracture
* Vitamin D levels < 30 ng/ml
* Patients with available medical history before and after initiation of study treatment
* Patients providing informed consent for this study

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patients receiving different osteoporosis treatment
* Patients with known hypersensitivity to vitamin D
* Patients participating in another similar study at the same time with other drugs
* Patients with vitamin D contraindications according to the medical instructions for use
* Patients with a fracture due to a traffic accident

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years of age with a low energy fracture will be included in the study.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-03-11 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Vitamin D levels of the patients after receiving vitamin D supplementation | 1 month, 3 months, 6 months and 12 months
  Measurement of 25(OH)D vitamin
Evaluation of BMD of the patients after receiving vitamin D supplementation | 12 months
  Measurement of Bone Mineral Density

SECONDARY OUTCOMES:
PTH | 1 month, 3 months, 6 months and 12 months
  Measurement of blood test of Parathyroid Hormone
TSH | 1 month, 3 months, 6 months and 12 months
  Measurement of blood test of Thyroid-stimulating Hormone
Ca | 1 month, 3 months, 6 months and 12 months
  Measurement of blood test of Calcium levels
P | 1 month, 3 months, 6 months and 12 months
  Measurement of blood test of Phosphorus levels
ALP | 1 month, 3 months, 6 months and 12 months
  Measurement of blood test of Alkaline phosphatase levels
Al | 1 month, 3 months, 6 months and 12 months
  Measurement of blood test of Albumin levels
Mg | 1 month, 3 months, 6 months and 12 months
  Measurement of blood test of Magnesium levels

CONTACTS AND LOCATIONS:
Locations (1):
- KAT General Hospital of Attika, Kifissia, Attica, Greece